CLINICAL TRIAL: NCT01026584
Title: Efficacy and Safety of Aripiprazole in Patients With First Episode Psychosis: an Open-label, Prospective Multi-center Study
Brief Title: Efficacy and Safety of Aripiprazole in First Episode Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBIRB0909-97
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: First Episode Psychosis
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- drug (Other)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 6 week prospective study

SUMMARY:
The aim of the study is to investigate the efficacy and safety of aripiprazole in patients with first episode psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-59 years and meet DSM-IV diagnostic criteria for first episode of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder NOS as assessed by using the Structured Clinical Interview for DSM-IV, research version.

Exclusion Criteria:

* Meeting DSM-IV criteria for another axis I diagnosis, including substance abuse or dependence
* Needing another nonantipsychotic psychotropic medication at enrollment
* Having a serious or unstable medical illness.
* Pregnant or lactating women or women without adequate contraception will be also excluded.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Symptoms assessment by objective rating scales | week 1
  PANSS total score, SANS, CGI
Symptoms assessment by objective rating scales | week 2
  PANSS total score, SANS, CGI
Symptoms assessment by objective rating scales | week 3
  PANSS total score, SANS, CGI
Symptoms assessment by objective rating scales | week 4
  PANSS total score, SANS, CGI
Symptoms assessment by objective rating scales | week 6
  PANSS total score, SANS, CGI

SECONDARY OUTCOMES:
Assessment of adverse events by objective rating scales and self report scales | week 1
  NIDSS(Neuroleptic induced deficit syndrome scale), BAS, SAS
Assessment of adverse events by objective rating scales and self report scales | week 2
  NIDSS(Neuroleptic induced deficit syndrome scale), BAS, SAS
Assessment of adverse events by objective rating scales and self report scales | week 4
  NIDSS(Neuroleptic induced deficit syndrome scale), BAS, SAS, AIMS
Assessment of adverse events by objective rating scales and self report scales | week 6
  NIDSS(Neuroleptic induced deficit syndrome scale), BAS, SAS, AIMS, Lipid profile

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Department of Psychiatry, Kangwon National University College of Medicine, Chunchon
  - Department of Psychiatry, Kyungpook national University School of Medicine, Daegu
  - Department of Psychiatry, Eulji University, School of Medicine, Daejeon
  - Department of Psychiatry, Kongju National Hospital, Gongju
  - Department of Psychiatry, Inje University College of Medicine, Ilsan Paik Hospital, Goyang
  - Department of Psychiatry, Chonnam National University Medical School, Hwasun
  - Department of Psychiatry, College of Medicine, Won-Kwang University, Iksan
  - Department of Psychiatry, Gachon University of Medicine and Science, Incheon
  - Department of Psychiatry, Chonbuk national University Hospital, Jeonju
  - Department of Psychiatry, Myongji Hospital Kwandong Uni. college of Medicine, Koyang
  - St. John of God Neuropsychiatric Hospital, Kwangju
  - department of Neuropsychiatry. Dong-Eui University Medical Center, Pusan
  - Department of Neuropsychiatry, Soonchunhyang University Hospital, Seoul